CLINICAL TRIAL: NCT05617144
Title: Aromatherapy Protocol for Pain Reduction in Hospice Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Tamara Blanton, Student, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-SN-21-1090
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Pain
Keywords: hospice care
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Other: Aromatherapy treatment

INTERVENTIONS:
Other: Aromatherapy treatment — 60 minutes after pain medication administration primary investigator will turn on the diffuser (manufacture ScentSationals)and administer aromatherapy with a mixture of four drops of lavender and four drops of peppermint for 60 minutes.

SUMMARY:
The purpose of this study is to introduce aromatherapy with current pain medication protocols to see if it improves patient satisfaction and reduces pain in hospice care patients.

ELIGIBILITY:
Inclusion Criteria:

* currently on hospice at Seasons Assisted Living

Exclusion Criteria:

* pain level not 3/10 or higher

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-01-08 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction as assessed by the score on the Patient Satisfaction survey | end of study (7 days after baseline)
  This survey has 4 questions and each is scored from 1(strongly disagree) to 5(strongly agree) for a maximum score of 20, a higher score indicating more satisfaction

SECONDARY OUTCOMES:
Change in pain as assessed by the score on the Wong Baker Face Scale (WBFPS) scale | Baseline, 2 hours after every aromatherapy administration
  This is scored from 0(no hurt) to 10(hurts the worst) a higher number indicating more pain

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Blanton, MS,RN, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No